# **RVT-1401-2003 Statistical Analysis Plan**

# Final Analysis – Cohort 1

Version 3.0

# **10 December 2021**

A Phase 2, Multicenter, Non-Randomized, Open Label Study of RVT-1401 for the Treatment of Patients with Warm Autoimmune Hemolytic Anemia Protocol (Version 3) Dated 23 December 2019

Immunovant Sciences GmbH
Viaduktstrasse 8
4051 Basel
Switzerland

#### CONFIDENTIALITY STATEMENT

This document contains confidential information. Any use, distribution, or disclosure without the prior written consent of Immunovant Sciences

GmbH is strictly prohibited except to the extent required under applicable laws or regulations. Persons to whom the information is disclosed

must be informed that the information is confidential and may not be further disclosed by them.

# TABLE OF CONTENTS

| TAB | LE OF CONTENTS | 2 |
|------|-------------------------------------------------|----|
| ABB | REVIATIONS | 4 |
| APP] | ROVAL | 6 |
| 1 1 | INTRODUCTION | 7 |
| 2 ( | OBJECTIVES AND ENDPOINTS | 7 |
| 2.1 | Objectives | 7 |
| 2.2 | Endpoints | 7 |
| 2. | 2.1 Primary Endpoints | 7 |
| 2. | 2.2 Secondary Endpoints | 7 |
| 2. | 2.3 Exploratory Endpoints | 8 |
| 3 5 | STUDY DESIGN | 8 |
| 3.1 | Sample Size and Statistical Power Consideration | 8 |
| 3.2 | Study Diagram and Flow Chart | 9 |
| 3.3 | Time and events table | 10 |
| 4 | ANALYSIS POPULATIONS (ANALYSIS SETS) | 14 |
| 4.1 | Efficacy Population | 14 |
| 4.2 | Safety Population | 14 |
| 4.3 | Pharmacokinetic Population | 14 |
| 4.4 | Pharmacodynamic Population | 14 |
| 5 | TREATMENT DESCRIPTIONS | 14 |
| 6 5 | STATISTICAL ANALYSIS METHODS AND ISSUES | 14 |
| 6.1 | Statistical Methods | 14 |
| 6.2 | Missing Data | 14 |

| 6.3 | Data Issues | 15 |
|------|---------------------------------------------------------|--------|
| 6.4 | Baseline Definition | 16 |
| 7 I | DISPOSITION, DEMOGRAPHICS AND BASELINE CHARACTERISTICS | 16 |
| 7.1 | Subject Disposition and Exposure | 16 |
| 7.2 | Demographics and Baseline Characteristics | 16 |
| 7.3 | Prior WAIHA treatment | 16 |
| 8 A | ANALYSIS OF EFFICACY ENDPOINTS | 16 |
| 9 A | ANALYSIS OF SAFETY ENDPOINTS | 17 |
| 9.1 | Adverse Events | 17 |
| 9.2 | Vital Signs | 17 |
| 9.3 | Laboratory Test Results | 17 |
| 9.3 | 3.1 Hematology | 17 |
| 9.3 | 3.2 Clinical Chemistry | 18 |
| 9.3 | 3.4 Lipid Panel | 18 |
| 9.4 | Concomitant Medications, Rescue Therapy, and Procedures | 19 |
| 9.5 | Electrocardiogram | 19 |
| 9.6 | Physical Examination. | 19 |
| 9.7 | Pregnancy Testing. | 19 |
| 9.8 | COVID-19 Impact | 19 |
| 10 A | ANALYSIS OF PHARMACOKINETIC, PHARMACODYNAMIC, AND ANT | T-DRUG |
| A | ANTIBODY ENDPOINTS | 19 |

#### **ABBREVIATIONS**

ADA Anti-drug antibody

ADCC Antibody dependent cell mediated cytotoxicity

AE Adverse event

AESI Adverse event of special interest
AIHA Autoimmune hemolytic anemia

ALT Alanine aminotransferase
AST Aspartate aminotransferase

ATC Anatomical Therapeutic Chemical

ATP Adult treatment panel
BMI Body mass index
BUN Blood urea nitrogen
CI Confidence intervals

CLL Chronic lymphocytic leukemia

CO<sub>2</sub> Carbon dioxide

CPK Serum creatine phosphokinase

CTCAE Common Terminology Criteria for Adverse Events

ECG Electrocardiogram

FSH Follicle stimulating hormone

GCP Good Clinical Practice

GGT Gamma glutamyl transferase

Hb Hemoglobin
HBV Hepatitis B virus
HCV Hepatitis C virus

HIV Human immunodeficiency virus

IB Investigator's brochure
ICF Informed consent form

ICH International conference on harmonization

IEC Independent ethics committee

IgAImmunoglobulin AIgGImmunoglobulin GIgMImmunoglobulin M

IND Investigational new drug
INR International normalized ratio


#### Dated 10 December 2021

IP Investigational product

IRB Institutional review board

ITP Idiopathic thrombocytopenia purpura

ITT Intent to treat

IUD Intrauterine device

LDH Lactic acid dehydrogenase

MCH Mean corpuscular hemoglobin

MCHC Mean corpuscular hemoglobin concentration

MCV Mean corpuscular volume

MedDRA Medical Dictionary for Drug Regulatory Activities

MRC Medical Research Council

PD Pharmacodynamics
PK Pharmacokinetics
RBC Red blood cell

SAP Statistical analysis plan

SGOT Serum glutamic-oxaloacetic transaminase SGPT Serum glutamic-pyruvic transaminase

TBL Total bilirubin

TEAE Treatment-emergent adverse event

WAIHA Warm Autoimmune Hemolytic Anemia

WBC White blood cell

WHO World Health Organization

Dated 10 December 2021

#### **APPROVAL**

# Authored and approved by



# Approved by



Dated 10 December 2021

#### 1 INTRODUCTION

This statistical analysis plan (SAP) contains the analysis information for the definition of the analysis populations, derivation of variables, convention of analysis scope, and statistical methodology for the analyses of safety and efficacy of RVT-1401 in the treatment of subjects with Warm Autoimmune Hemolytic Anemia (WAIHA). Based upon a composite review and data suggesting a drug-related effect of RVT-1401 on lipids, the study was paused, and a final analysis of Cohort 1 is being conducted based on the analyses outlined in this SAP. Subjects whose treatment was paused are referred to as curtailed.

At the time of the pause, 5 subjects had been enrolled in Cohort 1; 2 subjects completed the study through the Week 20 visit, 1 subject Early Terminated after Week 3, and 2 subjects were in the treatment period at the time of the pause. The analyses outlined in this plan pertain to the analysis of available data for Cohort 1.

The SAP Version 2.0 was created during the writing of the interim CSR for Cohort 1. A Sponsor decision was made to only include listings in the CSR given the small number of subjects, and SAP Version 2.0 reflects this decision.

This version of the SAP (Version 3.0) made further changes (such as removing all derived variables) to the SAP Version 2.0 to better align with the decision made to only include listings in the CSR.

#### 2 OBJECTIVES AND ENDPOINTS

# 2.1 Objectives

The objective of the study is to investigate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and efficacy of RVT-1401 (680 mg/weekly and 340 mg/weekly) in subjects with WAIHA.

# 2.2 Endpoints

#### 2.2.1 Primary Endpoints

The primary endpoints are as follows:

- The proportion of responders at Week 13 (defined as Hb level ≥10g/dL with at least a ≥2 g/dL increase from baseline without rescue therapy or blood transfusions in the previous two weeks).
- Assessment of safety and tolerability by analysis of adverse event (AE) data and changes from baseline in vital signs, ECGs, and clinical laboratory values.

#### 2.2.2 Secondary Endpoints

- Change from baseline in Hb levels,
- Time to response,
- Change from baseline in hematocrit levels,

Dated 10 December 2021

- Proportion of subjects with Hb levels in the normal range at Week 13,
- Time to achieving Hb levels in the normal range,
- Change from baseline in FACIT-F score,
- Change from baseline in Medical Research Council (MRC) breathlessness scale,
- Change from baseline in EQ-5D-3L score,
- Change from baseline in levels of total IgG & IgG subclasses (1-4),
- Concentration of RVT-1401 at pre-dose,
- Change from baseline in LDH, bilirubin, and haptoglobin, and
- Immunogenicity determined by change from pre-dose in anti-RVT-1401 antibodies, and characterization of any anti-RVT-1401 antibodies to confirm neutralization potential.

# 2.2.3 Exploratory Endpoints



#### 3 STUDY DESIGN

This is a Phase 2, non-randomized, sequential, open-label study to investigate the safety, tolerability, PK, PD, and efficacy of RVT-1401 (680 mg/weekly and 340 mg/weekly) in subjects with WAIHA. Two cohorts of subjects will be enrolled in a non-randomized sequential approach. Subjects will be enrolled into Cohort 1 (680 mg/weekly) first followed by Cohort 2 (340 mg/weekly). (See 5.2 Study Diagram and Flow Chart)

Following the initial dose at the Baseline Visit (Week 1, Day 1), study visits will occur weekly throughout the treatment period. Following the final dose at Week 12, visits will occur weekly through Week 14 and then at Week 16 and Week 20. Safety, PK, PD, and clinical assessments will be collected throughout the study.

# 3.1 Sample Size and Statistical Power Consideration

The sample size for this study was not determined using statistical methods. The sample size was chosen based on clinical and recruitment considerations for this Phase 2 study.

# 3.2 Study Diagram and Flow Chart



<sup>\*\*</sup>Note-Cohort 1 will enroll first followed by Cohort 2

Dated 10 December 2021

# 3.3 Time and events table

| | Screening <sup>1</sup> | | | | | | | ment Per<br>Weeks) | iod | | | | | | | -up Period<br>(eeks) | | Early<br>Withdrawal Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Timepoint<br>(Weeks) | Within 30 days | 1<br>(B/<br>L) | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 16 | 20 | |
| Time Window (days) | | | +/-1<br>day | +/-1<br>day | +/-1<br>day | +/-1<br>day | +/-1<br>Day | +/-1<br>day | +/-1<br>day | +/-1<br>day | +/-1<br>day | +/-1<br>day | +/-1<br>day | +/-2<br>days | +/-2<br>days | +/-2<br>days | +/-<br>2 days | |
| Informed consent | Х | | | | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | Х | Х | | | | | | | | | | | | | | | | |
| Demographics and medical history <sup>9</sup> | Х | | | | | | | | | | | | | | | | | |
| Height | Х | | | | | | | | | | | | | | | | | |
| Body weight | Х | Х | | | | | | | | | | | | | | | | |
| Complete physical examination | Х | Х | | | | | | | | | | | | | | | | |
| Brief physical examination | | | | | | | | | | | | | | | | | Х | Х |
| Vital signs <sup>2</sup> | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| 12-lead<br>Electrocardiogram <sup>2</sup> | Х | Х | | | Х | | | | Х | | | | Х | | | | Х | Х |
| Pregnancy test <sup>3</sup> (females) | Х | Х | Х | | Х | | Х | | Х | | Х | | Х | Х | | | Х | Х |
| Viral Serology | Х | | | | | | | | | | | | | | | | | |
| Vaccine Titers <sup>2</sup> | | Х | | | | | | | | | | | | Х | | | Х | Х |
| QuantiFERON® – TB<br>GOLD | Х | | | | | | | | | | | | | | | | | |
| Urinalysis <sup>2, 4</sup> | Х | Х | | Х | | Х | | Χ | | Х | | Х | | Х | | Х | Х | Х |
| Blood chemistry and hematology <sup>2, 8</sup> | Х | Х | Х | Х | Х | Х | | Х | | Х | | Х | | Х | Х | Х | Х | Х |
| Fasting Lipid Panel <sup>2</sup> | | Х | | | | | | | | | | | | Х | | | Х | Х |


Confidential

Dated 10 December 2021

| | Screening <sup>1</sup> | | Treatment Period<br>(Weeks) | | | | | | | | | Follow-<br>(W | Early<br>Withdrawal Visit | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Timepoint | Within 30 | 1 | | | | | | | | | | | | | | | | |
| (Weeks) | days | (B/<br>L) | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 16 | 20 | |
| | | | +/-1 | +/-1 | +/-1 | +/-1 | +/-1 | +/-1 | +/-1 | +/-1 | +/-1 | +/-1 | +/-1 | +/-2 | +/-2 | +/-2 | +/- | |
| Time Window (days) | | | day | day | day | day | Day | day | day | day | day | day | day | days | days | days | 2 days | |
| Serum complement<br>(CH50, C3) <sup>2</sup> | | Х | | Х | | Χ | | Χ | | Х | | Х | | Х | | Х | Х | Х |
| Immunoglobulins (IgM, IgA) <sup>2</sup> | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | Х | X |

| | Screening <sup>1</sup> | | | | | | | ment Per<br>Weeks) | iod | | | | | | | -up Period<br>eeks) | | Early<br>Withdrawal Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Timepoint<br>(Weeks) | Within 30<br>days | 1<br>(B/<br>L) | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 16 | 20 | |
| Time Window (days) | | | +/-1<br>day | +/-1<br>day | +/-1<br>day | +/-1<br>day | +/-1<br>Day | +/-1<br>day | +/-1<br>day | +/-1<br>day | +/-1<br>day | +/-1<br>day | +/-1<br>day | +/-2<br>days | +/-2<br>days | +/-2<br>days | +/-<br>2 days | |
| RVT-1401 PK sampling <sup>2</sup> | | Х | Х | Х | Х | Х | Х | | Х | | Х | | Х | Х | | | | Х |
| Total IgG <sup>2,6</sup> | Х | Х | Х | Х | Х | Х | Х | | Х | | Х | | Х | Х | Х | Х | Х | Х |
| Immunoglobins<br>(IgG subclasses) <sup>2</sup> | | Х | | Х | | | Х | | Х | | Х | | | Х | | Х | Х | X |
| Anti- RVT-<br>1401antibody <sup>2, 5</sup> | | Х | | Х | | Х | | | Х | | | | | Х | | | Х | Х |
| NAb Assessment <sup>2</sup> | | Х | | Х | | Х | | | Х | | | | | Х | | | Х | Х |
| Drug administration | ı | l X | X | l x | l x | l v | lv | X | l x | l x | l v | X | l x | | | | ı | |
| Drug administration | | | | | | Х | Х | | | | Х | | | | | | | |
| Injection Site Reaction <sup>7</sup> | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | | | | |
| FACIT-F Scale <sup>2</sup> | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | Х | X |
| MRC Breathlessness<br>Scale <sup>2</sup> | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | Х | Х |
| EQ-5D-3L <sup>2</sup> | | Х | | | | Х | | | | Х | | | | Х | | Х | Х | Х |
| Satisfaction<br>Questionnaire | | | | | | | | | | | | | | Х | | | | Х |
| Adverse events | Х | Χ | Χ | Х | Х | Х | Х | X | Х | Х | Х | Х | Х | X | Х | X | Х | Х |
| Concomitant medication | Х | Х | Х | X | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |


Screening can take place over multiple days.
 Assessments collected on dosing days will be collected pre-dose.

#### Dated 10 December 2021

- 3. Pregnancy tests will be collected pre-dose (via urine dipstick) on dosing days where specified. Serum pregnancy tests should be collected at screening and the final follow up visit.
- 4. Microalbumin/creatinine ratio at baseline, Week 13, and Week 20 only.
- 5. Subjects with treatment emergent positive results (change from baseline) for anti- RVT-1401 antibody at Week 20 will be requested to return at approximately 6-, 9-, and 12-months post-dose for additional samples or until their result is no longer positive. However, for purposes of safety follow-up and database lock participation ends at the Week 20 visit.
- 6. Two samples for IgG will be collected: one will be sent to the central lab for safety monitoring, while the other sample will be sent to Intertek as the PD endpoint.
- 7. Local injection site reactions will be assessed at approximately 10 minutes post dose.
- 8. Hematology, HbA1c and will be drawn for site local laboratory analysis, at minimum, and results collected in the instance where central laboratory samples are received hemolyzed. If other central laboratory tests are received hemolyzed, the local result will be captured in the eCRF.
- 9. History of WAIHA and prior WAIHA treatments will be captured in the eCRFs.

# 4 ANALYSIS POPULATIONS (ANALYSIS SETS)

The populations defined in this section guide the selection of subjects for a given set of listings.

# 4.1 Efficacy Population

All subjects who enroll in the study and receive at least one dose of study treatment and have a post-baseline visit will be included in the efficacy population.

# 4.2 Safety Population

All subjects who enroll in the study and receive at least one dose of study treatment will be included in the Safety Population. This will be the population for the safety analyses, as well as for presentation and summarization of baseline/demographic characteristics and subject disposition.

# 4.3 Pharmacokinetic Population

The PK Population will include all subjects who undergo PK sampling and have evaluable concentration-time data for analysis.

# 4.4 Pharmacodynamic Population

The PD population will include all subjects who have a baseline measure, along with a post baseline measure and receive at least one dose of study treatment.

#### 5 TREATMENT DESCRIPTIONS

Unless otherwise indicated, the treatment will be identified by RVT-1401 680 mg/week (Cohort 1).

#### 6 STATISTICAL ANALYSIS METHODS AND ISSUES

#### **6.1 Statistical Methods**

All available data will be presented in the data listings.

# **6.2** Missing Data

Other than missing dates as described below, no imputation methods will be used for missing data.

#### Missing dates are imputed in the following cases:

For the analysis of safety variables, only partial dates may be imputed; otherwise, missing data will be treated simply as missing. The algorithms for imputation of partial dates depend upon the parameter.

Adverse Event Onset

• If onset date is completely missing, date is set to date of first dose. If onset time is missing, the time will not be imputed.

- If year is present and month and day are missing or year and day are present and month is missing:
  - If year = year of first dose, then set month and day to month and day of first dose.
  - If year < year of first dose, then set month and day to December 31.
  - If year > year of first dose, then set month and day to January 1.
- If month and year are present and day is missing:
  - If year = year of first dose and
    - month = month of first dose, then set day to day of first dose date.
    - month < month of first dose, then set day to last day of month.
- For all other cases, set date to date of first dose.

#### Adverse Event End Date

- If year is present and month and day are missing or year and day are present and month is missing, set end month and day to December 31.
- If month and year are present and day is missing, set the day to last day of the month.
  - If fatal event, date is set to minimum of imputed end date and death date.
  - For all other cases, set date to missing.

The imputed dates must be logical, ensuring that no end date is after database lock or death or before the start date.

If site queries fail to resolve partial dates for laboratory values and vital signs, the date is missing and will not be imputed.

#### **6.3** Data Issues

Unless otherwise noted, values reported as greater than or less than some quantifiable limit (e.g., <1.0) will include the sign in all listings.

If there are multiple assessments collected on the same scheduled time, all values will be displayed. All data from all visits will be eligible for inclusion in the listings.

Study day is the day relative to the date of first dose. Day 1 is defined as the date of first dose, unless otherwise specified for the calculation of baseline.

For visits (or events) after first dose, day is calculated as:

• Study day = visit (or event) date - date of first dose + 1

For visits (or events) before first dose, day is calculated as:

• Study day = visit (or event) date - date of first dose

Dated 10 December 2021

#### **6.4** Baseline Definition

Baseline is the last available assessment prior to time of the first dose unless it is specified otherwise.

Subject's age in years at baseline is defined as the age derived at Screening in the EDC system.

# 7 DISPOSITION, DEMOGRAPHICS AND BASELINE CHARACTERISTICS

# 7.1 Subject Disposition and Exposure

The disposition listing will include the disposition of treatment and discontinuation of study by each subject. For discontinuations, the listing will include the reason for discontinuation.

Disposition of subjects in the Follow-up Period will be presented in listings.

Administration of RVT-1401 will be presented in listings denoting each visit and dose, and the treatment satisfaction questionnaire will be listed by treatment and by visit.

WAIHA treatment listing will also be provided.

# 7.2 Demographics and Baseline Characteristics

The demographics (age, gender, race, ethnicity, and childbearing potential if female) and baseline characteristics (height, weight, body mass index) will be presented in listings.

#### 7.3 Prior WAIHA treatment

Based on the coded data of prior WAIHA medication(s) using the World Health Organization (WHO) Drug Reference List, the data will be presented in listings per the Anatomical Therapeutic Chemical (ATC) classification.

#### 8 ANALYSIS OF EFFICACY ENDPOINTS

Each endpoint noted below will be presented in a listing.

- FACIT-F score
- MRC breathlessness scale
- EQ-5D-3L score



#### 9 ANALYSIS OF SAFETY ENDPOINTS

Safety analyses will be performed on the Safety population unless otherwise indicated.

#### 9.1 Adverse Events

The adverse events (AEs) will be coded by the Medical Dictionary for Drug Regulatory Activities (MedDRA) version 22.1 or higher. A treatment-emergent adverse event (TEAE) is defined as any AE onset post first treatment. A listing of all subjects reporting TEAEs will be presented. A separate listing of serious TEAEs will be provided. A by-subject listing containing the AEs by the MedDRA system organ class and preferred term will be created. This listing will include start and end dates of the event, severity, and relationship to study drug. Injection site reactions will also be presented in a separate listing.

The AE data will not be imputed other than a missing date.

# 9.2 Vital Signs

The vital signs (systolic / diastolic blood pressure, pulse rate, pulse oximetry, and body temperature) will be presented in a listing at each visit.

# 9.3 Laboratory Test Results

The test results of clinical chemistry, hematology, and urinalysis (including the lipid panel) are to be presented in listings by visit.

All test results will be presented in listings.

#### 9.3.1 Hematology

| Platelet Count: | RBC Indices: | Automated WBC Differential: |
|---|---|---|
| Red Blood Cell (RBC) Count | Mean corpuscular volume (MCV) | Neutrophils |
| White Blood Cell (WBC) Count (absolute) | Mean corpuscular<br>hemoglobin<br>(MCH) | Lymphocytes |
| Reticulocyte Count | Mean corpuscular hemoglobin concentration (MCHC) | Monocytes |
| Hemoglobin | | Eosinophils |
| Hematocrit | | Basophils |
| Haptoglobin | | |

#### 9.3.2 Clinical Chemistry

| Blood urea<br>nitrogen (BUN) | Potassium | AST (SGOT) | Total (TBL)<br>and direct<br>bilirubin |
|---|---|---|---|
| Creatinine | Chloride | ALT (SGPT) | Uric Acid |
| Total Protein | Total carbon dioxide (CO <sub>2</sub> ) | Gamma glutamyl transferase (GGT) | Albumin |
| Sodium | Calcium (corrected) | Alkaline phosphatase (ALP) | Lactic acid<br>dehydrogenase<br>(LDH) |
| Serum<br>complement<br>(CH50, C3) | Immunoglobulin<br>M (IgM) | Immunoglobulin<br>A (IgA) | Immunoglobulin<br>G (IgG) |
| HbA1c | | | |

## 9.3.3 Routine Urinalysis

- Specific gravity, pH
- Glucose, protein, blood, and ketones by dipstick
- Microscopic examination (if blood or urine protein is abnormal)
- Microalbumin/creatinine ratio at baseline, Week 12, and Week 20, only if urine protein is abnormal

#### 9.3.4 Lipid Panel

- Total cholesterol
- HDL cholesterol
- LDL cholesterol (calculated)
- Non-HDL cholesterol (calculated)
- Triglycerides
- Total cholesterol/HDL cholesterol ratio (calculated)
- LDL / HDL cholesterol ratio (calculated)

Analyses will include the following:

- Listings of raw lipid values will be provided.
- Listings for the full lipid panel will be presented.

# 9.4 Concomitant Medications, Rescue Therapy, and Procedures

Based on the coded data of concomitant medication using the WHO Drug Reference List, the concomitant medications and rescue therapy will be presented in a listing per the ATC classification.

Procedures will be listed by treatment and by subject.

# 9.5 Electrocardiogram

The parameters of electrocardiography will be presented in a listing by visit. The overall evaluation (Normal/Abnormal) will be included as well.

# 9.6 Physical Examination

Physical examination listing will be provided by treatment and by visit.

# 9.7 Pregnancy Testing

Pregnancy testing will be listed by treatment and by visit.

# 9.8 COVID-19 Impact

COVID-19 impact on study visits and the reason for impact will be listed by treatment and by visit.

COVID-19 impact on study and treatment discontinuation will be listed by treatment and by visit.

# 10 ANALYSIS OF PHARMACOKINETIC, PHARMACODYNAMIC, AND ANTI-DRUG ANTIBODY ENDPOINTS

- Serum total IgG concentrations will be listed by subject and visit and will include treatment, date and time of sample collection, and the actual time (days) that the PD sample was collected relative to the prior dose.
- Serum RVT-1401 concentrations will be listed by subject and visit and will include treatment, date and time of sample collection, and the actual time (days) that the PK sample was collected relative to the prior dose.

Anti-drug antibody results will be listed by subject and visit and will include treatment and date and time of sample collection.

#### **Certificate Of Completion**

Envelope Id: 78AD8323967C4CE993A140AAA427953D

Subject: Please DocuSign: Immunovant\_RVT-1401-2003 v3.0 SAP.docx

Source Envelope:

Document Pages: 19 Certificate Pages: 5

AutoNav: Enabled

Envelopeld Stamping: Disabled

Time Zone: (UTC-08:00) Pacific Time (US & Canada)

Status: Completed

Envelope Originator:



Sent: 12/10/2021 8:44:34 AM Viewed: 12/13/2021 11:19:17 AM Signed: 12/13/2021 11:19:52 AM

Sent: 12/10/2021 8:44:33 AM Viewed: 12/10/2021 8:44:47 AM

Signed: 12/10/2021 8:45:06 AM

IP Address:

#### **Record Tracking**

Status: Original

12/10/2021 8:41:20 AM

Holder:

Location: DocuSign

**Timestamp** 

#### **Signer Events**

**Immunovant** 

Security Level: Email, Account Authentication (Required)

Signature

Signatures: 2

Initials: 0



Signature Adoption: Pre-selected Style

Signature ID:

Using IP Address:

With Signing Authentication via DocuSign password With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 8/12/2021 6:15:18 AM ID: 1ff0aca2-79b9-439e-b7fd-c714265caa3d



Security Level: Email, Account Authentication

(Required)



Signature Adoption: Pre-selected Style

Signature ID:

Using IP Address:

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

#### **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

| In Person Signer Events | Signature | Timestamp |
|------------------------------|-----------|-----------|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |

| Carbon Copy Events | Status | Timestamp |
|---|---|---|
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 12/10/2021 8:44:34 AM |
| Certified Delivered | Security Checked | 12/10/2021 8:44:47 AM |
| Signing Complete | Security Checked | 12/10/2021 8:45:06 AM |
| Completed | Security Checked | 12/13/2021 11:19:52 AM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, SHI OBO Immunovant, Inc. - GxP Compliant Part 11 (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

# Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

## How to contact SHI OBO Immunovant, Inc. - GxP Compliant Part 11:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to:

#### To advise SHI OBO Immunovant, Inc. - GxP Compliant Part 11 of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

#### To request paper copies from SHI OBO Immunovant, Inc. - GxP Compliant Part 11

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to an email to an email to an email to be an email and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with SHI OBO Immunovant, Inc. - GxP Compliant Part 11

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to an and in the body of such request you must state your email, full name, mailing address, and telephone number. Reason for withdrawing consent. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process.

#### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

#### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify SHI OBO Immunovant, Inc. GxP Compliant Part 11 as
  described above, you consent to receive exclusively through electronic means all notices,
  disclosures, authorizations, acknowledgements, and other documents that are required to
  be provided or made available to you by SHI OBO Immunovant, Inc. GxP Compliant
  Part 11 during the course of your relationship with SHI OBO Immunovant, Inc. GxP
  Compliant Part 11.